CLINICAL TRIAL: NCT06802120
Title: Effects of Osteopathic Management on Disability and Quality of Life After Lumbar Arthrodesis. A PARALLEL, RANDOMIZED AND DOUBLE-BLIND CONTROLLED PILOT STUDY
Brief Title: Effects of Osteopathic Management on Disability and Quality of Life After Lumbar Arthrodesis
Acronym: OSTEODESE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Bizet (Other)
Collaborators: Institut De La Colonne Vertebrale Et Des Neurosciences (Other); Ecole Supérieur d'Ostéopathie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2024-A01768-39
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Chirurgical Intervention

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted osteopathic treatment (Experimental): treatment with real osteopathy
  Interventions: Other: osteopathy real
- Non-targeted osteopathic treatment (Placebo Comparator): treatment with sham osteopathy
  Interventions: Other: sham osteopathy

INTERVENTIONS:
Other: osteopathy real — treatment with real osteopathy 2 times a week for 8 weeks
  Arms: Targeted osteopathic treatment
Other: sham osteopathy — treatment with sham osteopathy 2 times a week for 8 weeks
  Arms: Non-targeted osteopathic treatment

SUMMARY:
The aim of our study is to assess the effect of a combined physiotherapy and osteopathy treatment versus a placebo on the management of disability and quality of life after lumbar arthrodesis. This study will provide a better assessment of the use of osteopathy as a non pharmacological approach to post-operative management.

For this purpose, We will analyze the effects of these two approaches, targeted and non-targeted osteopathy (TO vs. NTO), on patients' disability and quality of life after surgery.

ELIGIBILITY:
Inclusion Criteria:

* having experienced a lumbar arthrodesis (of one to three levels) four weeks before inclusion
* being under a stable pharmacological treatment over the last month
* who are suffering from postoperative mechanical pain (VAS ≥ 4)

Exclusion Criteria:

* neuropathic pain according to a DN4 score greater than or equal to 4/10,
* are suffering from fibromyalgia,
* algodystrophy,
* other somatic or neuropsychiatric diseases (other than depression and anxiety),
* have received osteopathic treatment over the last three month prior to inclusion,
* are included in another interventional research protocol during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Disability will be assessed using the ODQ | baseline and Week 8
  Oswestry Low Back Pain Disability Questionnaire
  * Minimum Value: 0
  * Maximum Value: 100
  * Interpretation: Higher scores indicate a worse outcome => greater disability due to low back pain.

SECONDARY OUTCOMES:
Pain and disability measures | baseline, ans every week from 1 to 8
  The Visual Analog Scale is a subjective measurement tool commonly used to assess the intensity of pain. It consists of a horizontal 10-centimeter line on which the patient marks a point that reflects their experience. Minimum and maximum values: 0 = complete absence of the symptom 10 = the most severe imaginable intensity of the symptom Score interpretation: Higher scores indicate greater symptom intensity Lower scores indicate lesser intensity
The Osteopathic Dysfunction Palpation Assessment Scale | baseline and Week 8
  Osteopathic Dysfunction Palpation Assessment Scale
  Minimum value: 0 (no dysfunction detected)
  Maximum value:
  Each anatomical structure (e.g., ilium, pubis, sacrum, spine, etc.) is assessed on 4 criteria: mobility, viscoelasticity, texture, temperature.
  For each criterion, the score is 0 or 1 (absence or presence of dysfunction). For each structure, the maximum score is therefore 4. The total maximum score depends on the number of structures assessed
  Interpretation: The higher the score, the greater the osteopathic dysfunction (so a higher score indicates a worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Bizet, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided